CLINICAL TRIAL: NCT06488976
Title: Development of a New Scoring System for Enuresis Nocturna: Nocturnal Enuresis Symptom Score (NESS)
Brief Title: Nocturnal Enuresis Symptom Score
Acronym: NESS
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tarik Emre Sener, Associating Professor, MD, Marmara University
Other Study IDs: MAR.UAD.010
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Enuresis, Nocturnal
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Enuresis nocturna: Patients older than 5 years of age and the main compliment should be bedwetting without any history of additional lower urinary tract symptoms.
- Healthy control: Patients older than 5 years of age, no remarkable past medical history and complaints.

SUMMARY:
Monosymptomatic nocturnal enuresis (NE), also known as bedwetting, is also defined as intermittent nocturnal enuresis.

Nocturnal enuresis is considered primary when a child has not yet been dry for an extended period of time (six months). The term "secondary NE" is used when a child or adult starts wetting again after being dry for at least 6 months.

Non-monosymptomatic NE is used for patients with lower urinary tract-related voiding symptoms (frequent urination, intermittent voiding, incomplete voiding, urinary tract infection, sudden urge to urinate during the daytime, daytime urinary incontinence).

It is a relatively common symptom in children, with an incidence of 5-10% at the age of seven and 1-2% in adolescents. The ratio of girls to boys has been reported in the literature as roughly 2 to 1.

The annual spontaneous resolution rate is 15% (at any age) and it is considered a relatively benign condition.

Enuresis nocturne has important secondary stressful, emotional and social consequences for children.

Caregivers (caregivers, parents, etc.) of these patients have reported a lower quality of life compared to control groups in studies.

Since children under 5 years of age have a very high probability of spontaneous resolution, the European Society of Urology Guidelines recommend treating children over 5 years of age.

Seven out of 100 seven-year-old bedwetting children will continue to wet the bed in adulthood.

Initially, conservative methods should be recommended, supportive measures including normal and regular eating and drinking habits should be planned, fluid intake should be restricted 3 hours before bedtime and urination should be encouraged by going to the toilet before going to bed at night.

In cases where conservative treatment fails to elicit a response, the child is awakened at a planned time at night with alarm therapy and taken to the toilet to urinate. Thus, it is aimed to empty the urine in the bladder and prevent bedwetting, but with this method, the sleep quality of the child and caregiver is shaken and the quality of life is reduced.

Another treatment method is sublingual desmopressin administration as a medical treatment. The dose frequently used in children has been reported as 120 mcg/day and found to be safe.

In case of dose inadequacy or inadequate response, there are reports showing that 240 mcg desmopressin sublingual treatment is also effective and safe.

Despite sequential and combined treatments, inadequate treatment response may occur in 10-15% of patients or bedwetting symptoms may recur in 25-30% of patients after treatment. In these patients, invasive examinations such as urodynamics and cystoscopy may be planned if necessary, depending on the results of the review after a detailed lower urinary tract function questioning.

There is no questionnaire for primary monosymptomatic enuresis nocturna in the literature. This makes categorization of patients, differential diagnosis, treatment monitoring and response evaluation difficult.

Our aim with this study is that this form will play an active role in categorizing patients and choosing between different treatment modalities at the diagnosis and treatment monitoring stages and will be a helpful tool for clinicians in the future.

DETAILED DESCRIPTION:
Primary monsymptomatic enuresis nocturna is defined as unrecognized urinary incontinence at night in children under the age of 18 years and over the age of 5 years, but it is essential to understand that there are no daytime symptoms or voiding symptoms in this disease. In this context, uroflowmetry, residual urine measurement, voiding dysfunction symptom score (VDSS), bladder diary and urinalysis are frequently used in the evaluation of lower urinary tract symptoms in the diagnosis and follow-up stages.

In this clinical study, a symptom questionnaire form will be filled out by asking the relatives and participants with primary monosymptomatic enuresis nocturna who will be admitted to the pediatric urology outpatient clinic between 15.01.2024-15.10.2024. The data and questionnaire results of the first 20 patients (healthy and volunteer) and the reliability and validity of the questionnaire will be statistically evaluated with Cronbach's alpha method and the number of patients will be completed to 200 after the reliability of the questionnaire is completed with this pilot study. Volunteer (healthy) patients will not undergo any additional examination/testing/treatment within the study, except for the physical examination performed in the routine pediatric urology outpatient clinic.

The reason for including healthy volunteers in the study was to measure whether the questionnaire would also be negative in patients who did not complain of nighttime bedwetting. This questionnaire consists of 9 questions in Turkish language and it is planned to mark only one answer per question for each patient. Total scores and answers given per question will be evaluated separately. The results of the tests ordered by our outpatient clinic from patients with a diagnosis of enuresis nocturna will be evaluated by the faculty members of Department of Urology and Division of Pediatric Urology, voiding flow curves and urine volume measurements remaining in the bladder after voiding, frequency-volume measurements in bladder diaries, The severity of enuresis nocturna will be evaluated by noting voiding dysfunction symptom scores (VDSS), renal function tests, complete urine tests, physical examination findings and standard treatments in accordance with the literature and guidelines will be applied (alarm therapy, conservative approaches and desmopressin therapy). It will be investigated whether the scores generated by the forms will be helpful in predicting treatment response and selection. Patients who will be included in the study will not require a re-examination or additional examination/treatment, and no non-standard evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of primary and monosymptomatic enuresis nocturna.

Exclusion Criteria:

* Patients with a known urogenital anatomical disorder
* Patients with an additional one lower urinary tract symptom
* Patients that been dry at the nights for >6 months in any time period over the age of 5.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients with primary monosymptomatic enuresis nocturna who will be admitted to the pediatric urology outpatient clinic of our center between 15.01.2024-15.10.2024.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-10-26 (Actual)

PRIMARY OUTCOMES:
Internal consistency of questionnarre | 15.01.2024-01.08.2024
  Form will be analysed by Cronbach's alpha.
External validation of questionnarre | 15.01.2024-01.08.2024
  Form will be applied to another patient population

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, School of Medicince, Department of Urology, Pediatric Urology Division, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided